CLINICAL TRIAL: NCT03106818
Title: Postoperative Pain Alleviation in Patients Undergoing Cardiac Surgery; Presternal Bupivacaine and Magnesium Infiltration Versus Conventional Intravenous Analgesia
Brief Title: Postoperative Pain Alleviation in Open Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, lecturer of anesthesia and ICU, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00009911
Record Dates: First submitted 2017-04-04; First posted 2017-04-10 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Open Heart Surgery; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Magnesium Sulfate; Anesthetics, Local; Adjuvants, Pharmaceutic; Congresses as Topic; Acetaminophen; Ketorolac

STUDY DESIGN:
Intervention Model Description: pain control in the early postoperative period
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A (Active Comparator): ( bupivacain 0.125% magnesium sulfate 5%) infusion in the presternum , for 48 hours
  Interventions: Drug: bupivacain with magnesium sulphate
- group B (Active Comparator): bupivacaine 0.125% infusion in the presternum , for 48 hours
  Interventions: Drug: Bupivacaine only
- Group C (Active Comparator): will be conventional , will receive postoperative fentanyl , paracetamol , and ketorolac.
  Interventions: Drug: conventional

INTERVENTIONS:
Drug: bupivacain with magnesium sulphate — will receive bupivacain 0.125% and magnesium sulphate 5% infusion in the presternum , for 48 hours
  Other Names: local anesthetic with adjuvant for 48 hours
  Arms: group A
Drug: Bupivacaine only — will receive bupivacain 0.125% infusion in the presternum , for 48 hours
  Other Names: local anesthetic
  Arms: group B
Drug: conventional — only conventional post operative analgesics will be used
  Other Names: paracetamol , Ketorolac
  Arms: Group C

SUMMARY:
Effective pain relief after cardiac surgery has assumed importance with the introduction of fast track discharge protocols that requires early weaning from mechanical ventilation. Inadequate pain control reduces the capacity to cough, mobility, increases the frequency of atelectasis, and prolongs recovery. Infiltration of local anesthetics near the surgical wound has shown to improve early postoperative pain in various surgical procedures.

Magnesium is the fourth most plentiful cation in our body. It has antinociceptive effects in animal and human models of pain.

DETAILED DESCRIPTION:
Effective pain relief after cardiac surgery has assumed importance with the introduction of fast track discharge protocols that requires early weaning from mechanical ventilation. Inadequate pain control reduces the capacity to cough, mobility, increases the frequency of atelectasis, and prolongs recovery.

A major cause of pain after cardiac surgery is the median sternotomy particularly on the first two postoperative days.

The most often used analgesics in these patients are parenteral opioids which can lead to undesirable side-effects as sedation, respiratory depression, nausea, and vomiting.

Infiltration of local anesthetics near the surgical wound has shown to improve early postoperative pain in various surgical procedures.

Magnesium is the fourth most plentiful cation in our body. It has antinociceptive effects in animal and human models of pain.

It has been mentioned in a systematic review that it may be worthwhile to further study the role of supplemental magnesium in providing perioperative analgesia, because this is a relatively harmless molecule, is not expensive and also because the biological basis for its potential antinociceptive effect is promising.

These effects are primarily based on physiological calcium antagonism, that is voltage-dependent regulation of calcium influx into the cell, and noncompetitive antagonism of N-methyl-D-aspartate (NMDA) receptors.

there is a need to evaluate and compare local magnesium with bupivacaine , in comparison to bupivacain ,and other conventional intarvenous analgesics

ELIGIBILITY:
Criteria:

Inclusion Criteria:

* 18-60 years old
* American Society of Anesthesiologists physical status II and III
* Patients scheduled for open heart valve replacement surgery with sternotomy

Exclusion Criteria:

* Emergency surgery
* Clinically significant kidney or liver disease
* Patients allergic to local anesthetic
* Patients with prolonged CPB time (>120 min)
* Patients required intra-aortic balloon pump

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
postoperative pain | 48 hours postoperative
  Vas Scale

SECONDARY OUTCOMES:
extubation time | 48 hours
  time to separate patient from mechanical ventilation and extubation
Fentanyl consumption | 48 hours
  total fenatnyl consumption

CONTACTS AND LOCATIONS:
Overall Officials: Emad Kamel Said, MD, Principal Investigator — Anesthesia departement , Faculty of Medicine , Assiut university
Locations (1):
- Emad Zarief Kamel Said, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No